CLINICAL TRIAL: NCT02950389
Title: REmoval of Free Light Chains in Hemodialysis Patients Without Multiple Myeloma. A Crossover COmpaRison of Three Different dialyzERs
Brief Title: REmoval of Free Light Chains. A COmpaRison of Three Different dialyzERs
Acronym: RECORDER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Gabriele Donati, M.D. Ph.D., IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 2016/GD/2
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Complication of Hemodialysis
Keywords: PMMA; on-line HFR; free light chains; toxins; removal; hemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Six bicarbonate dialysis session with PMMA dialysis filter for 2 weeks, followed by 2 weeks of 6 on-line HFR session with HFR17 dialysis filter, than 6 bicarbonate dialysis session for 2 weeks with F7 dialysis filter.
  Interventions: Device: PMMA filter; Device: HFR17 filter; Device: F7 filter
- Group B (Experimental): Six on-line HFR session with HFR17 dialysis filter for 2 weeks, followed by 2 weeks of 6 o bicarbonate dialysis session with PMMA dialysis filter for 2 weeks, than 6 bicarbonate dialysis session for 2 weeks with F7 dialysis filter.
  Interventions: Device: PMMA filter; Device: HFR17 filter; Device: F7 filter

INTERVENTIONS:
Device: PMMA filter
Device: HFR17 filter
Device: F7 filter

SUMMARY:
Immunoglobulin light chains are classified as middle molecule uremic toxins able to interact with B lymphocyte membranes leading to the activation of transmembrane signaling. The ensuing impairment of neutrophil function can contribute to the chronic inflammation state of uremic patients, and the increased risk of bacterial infections or vascular calcifications. The aim of this crossover observational study was to assess the difference in free light chain removal by three different hemodialysis filters in patients not affected by multiple myeloma.

Free light chain removal was compared in the polymethylmethacrylate (PMMA) membrane Filtryzer BK-F, the polyphenylene HFR17 filter and the conventional polysulfone filter F7 High Performance dialysers (HPS). Twenty chronic hemodialysis patients were enrolled. The patients were randomized into two groups of treatment lasting six weeks each. The dialysis sessions checked were the midweek sessions and the blood was drawn at times 0, 120' and 240'. Kappa (k) and lambda (l) light chain levels, beta2microglobulin (β2M), C reactive protein (CRP) and albumin were checked.

DETAILED DESCRIPTION:
Background. Immunoglobulin light chains are classified as middle molecule uremic toxins together with β2M and parathyroid hormon. They have a mean molecular weight of 25,000 daltons for monomers (k free light chains) and approximately 50,000 daltons for dimers (lambda free light chains).

Raised serum levels of polyclonal free light chains can impair neutrophil function in terms of: 1) inhibited chemotactic movement; 2) reduced activation of glucose uptake; 3) inhibited apoptosis.

Immunoglobulin light chains are able to interact with B lymphocyte membranes leading to the activation of transmembrane signaling . The ensuing impairment of neutrophil function can contribute to the chronic inflammation state of uremic patients and to the increased risk of bacterial infection. Desjardins et al. demonstrated an association between free light chain levels and vascular calcification progression in chronic kidney disease patients. Nonetheless, serum free light chains in patients with chronic kidney disease are associated with the risk of end stage renal disease and death.

It seems that high flux PMMA membranes significantly reduce the light chain level, presumably due to adsorption. This behavior has led to the use of PMMA in the removal of monoclonal free light chains during multiple myeloma.

Preliminary reports describe a significant reduction in free light chains also during hemodiafiltration with reinfusion of endogenous ultrafiltrate (on-line HFR). A recent paper by Borrelli et al. reported an improvement in chronic inflammation after chronic online HFR in dialysis patients.

The aim of this crossover observational study was to compare free light chain removal by three different hemodialysis filters in a cohort of chronic dialysis patients not affected by multiple myeloma.

Methods. One hundred and sixty-three patients on chronic hemodialysis at the Nephrology, Dialysis and Transplantation Unit of S.Orsola University Hospital in Bologna were considered for the study.

The inclusion criteria were free light chain values >100 mg/L for k chains and >50 mg/L for lambda chains. These levels were chosen arbitrarily because no cut-off levels are available in the literature for the assessment of lowered serum free light chain values during hemodialysis in patients with end-stage renal disease. Other inclusion criteria were: age >18 years, absence or <200 ml/die residual diuresis, fistula or central venous catheter with blood flow >250 ml/min. Exclusion criteria were: intradialytic hypotension during bicarbonate dialysis, multiple myeloma requiring the double PMMA filter application, poly-allergy, HIV positivity. The filters used during the study were: i) HFR17 (Bellco, Mirandola, Italy), a double chamber filter used for online HFR. The first part of the filter consisted in a polyphenylene high flux hemofilter with an ultrafiltration coefficient (Kuf) of 28 ml/h/mmHg, a surface area of 0.7 m2 and a membrane cut-off value of 35,000 daltons. The endogenous ultrafiltrate rate is obtained automatically by means of the transmembrane pressure levels in the hemofilter. These are calculated from two pressure sensors: the first is on the arterial bubble chamber and the second before the roller pump of the ultrafiltrate. The ultrafiltrate is driven from this hemofilter to a 40 g neutral styrenic resin that allows an adsorbing area of 28,000 m2. After adsorption, the ultrafiltrate is added to the whole blood that, in turn, passes into the second HFR17 filter, a polyphenylene low flux filter (Kuf 13 ml/h/mmHg, surface area 1.7 m2) where the weight loss and diffusive depuration take place. ii) PMMA (Toray Filtryzer BK-F, Tokyo, Japan) with a surface area of 2.1 m2, a membrane cut-off value of 20,000 daltons and an ultrafiltration coefficient (Kuf) of 26 ml/h/mmHg. iii) A conventional polysulfone membrane (Fresenius F7HPS, Bad Homburg, Germany) with a cut-off of 11,500 daltons, a Kuf of 16 ml/h/mmHg and a surface area of 1.7 m2 was used as a control dialyzer.

The patients enrolled were randomized into two groups of treatments lasting six weeks each. Group A: 1st and 2nd weeks with bicarbonate dialysis and filter PMMA, 3rd and 4th weeks with filter HFR17, 5th and 6th weeks with bicarbonate dialysis filter F7. Group B: 1st and 2nd weeks with filter HFR17, 3rd and 4th weeks with bicarbonate dialysis and filter PMMA, 5th and 6th weeks with bicarbonate dialysis filter F7. The dialysis sessions carried out during weeks 1, 3 and 5 were considered washout sessions between weeks 2, 4 and 6 when the assessment of lambda and k light chains, β2M, C reactive protein and albumin was scheduled. Week number 1 was the washout period between the usual dialytic treatment of the patients enrolled and the beginning of the study. The checking dialysis session was the midweek session and the blood was drawn on starting dialysis (time 0), at two hours (time 120') and at dialysis end (time 240'). All the dialysis sessions lasted four hours. Mean blood flow was 310±30 ml/min, the mean ultrafiltration rate was 700±200 ml/h, during HFR the endogenous ultrafiltrate rate was 2.3±0.4 ml/h. Dialysate flow was 500 ml/min. Low molecular weight heparin enoxaparin (Clexane®, Sanofi, Milan, Italy) was used for anticoagulation of the extracorporeal circuit. Doses of 2000 IU (patients <50 kg of body weight), 4000 IU (patients between 50 to 90 kg of body weight) or 6000 IU (patients >90 kg of body weight) were administered in a single bolus on starting dialysis. Fresenius 5008 and Bellco Flexya dialysis machines were used. The concentrations of k and lambda light chains and β2M were measured by nephelometry (kit Freelite k/lambda, The Binding Site Group Ltd., Birmingham, United Kingdom; IIMAGE/IMMAGE 800 Beckman Coulter instrument, Brea California USA, Beckman Coulter β2M kit). Normal values: k light chains 3.3 -19.9 mg/L, lambda light chains 5.7-26.3 mg/L, β2M 0.7 - 2 mg/L. Molecular weights: k light chains: 22,500 daltons; lambda light chains: 45,000 daltons; β2M: 11,818 daltons. The reference range for patients with normal kidney function was considered between 0.26 and 1.65 according to Bourguignon et al.. CRP concentration was measured by turbidimetry (CRPLX, Tina-quant C-Reactive-Protein; Roche/Hitachi 902 analyzer). CRP normal value < 0.8 mg/dl, molecular weight 120,000 daltons. Albumin was assessed using the common laboratory method. The reduction rate per session (RRs) was calculated as follows:

RRs = (Cpre- Cpost-corr)/ Cpre x 100 (1) where Cpre is the predialysis solute level, and Cpost-corr is the post-dialysis solute concentration. The values measured during dialysis were corrected for hemoconcentration due to the patient's weight loss assuming a unicompartmental behavior of light chains described by the following formula: Cpost-corr = Cpost/ {1+ [DeltaBW/(0.2xBWpost)]} (2) where Cpost-corr is the post-dialysis solute concentration and Cpost-corr is the concentration of light chains corrected for the hemoconcentration, Delta body weight (DeltaBW) is the weight subtracted during dialysis, and BW (body weight) is the body weight at the end of dialysis.

Statistical analyses. Statistical analysis was performed using the "Statistical package for the social sciences (SPSS)" statistical software. The data are presented as mean ± standard error of the mean. The Shapiro-Wilk test, suitable for small populations, showed a non-normal distribution of the variables, for which the non-parametric Friedman test was used. The p value <0.05 was considered normal. The Wilcoxon Signed Rank Test was subsequently used to see which pairwise comparisons resulted statistically different. In addition, as a multiple comparison was done, we applied the Bonferroni correction, thereby setting a p value = 0.05 / 3 = 0.0167. For each of the sampling times 0.120 and 240 minutes, we compared the results and the RRs obtained with the different filters (HFR17, PMMA, F7).

ELIGIBILITY:
Inclusion Criteria:

* chronic hemodialysis patients
* free light chain values >100 mg/L for k chains or >50 mg/L for lambda chains.
* absence or <200 ml/die residual diuresis
* fistula or central venous catheter with blood flow >250 ml/min.

Exclusion Criteria:

* intradialytic hypotension
* multiple myeloma
* poly-allergy
* HIV positivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Compare free light chain removal by three different hemodialysis filters in a cohort of chronic dialysis patients not affected by multiple myeloma | 45 days

SECONDARY OUTCOMES:
Compare beta 2 microglobulin removal by three different hemodialysis filters | 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Donati, MD, PhD, Principal Investigator — S.Orsola University Hospital, Nephrology Dialysis and Renal Transplantation Unit
Locations (1):
- Nephrology Dialysis and Renal Transplantation Unit, S.Orsola University Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vanholder R, De Smet R, Glorieux G, Argiles A, Baurmeister U, Brunet P, Clark W, Cohen G, De Deyn PP, Deppisch R, Descamps-Latscha B, Henle T, Jorres A, Lemke HD, Massy ZA, Passlick-Deetjen J, Rodriguez M, Stegmayr B, Stenvinkel P, Tetta C, Wanner C, Zidek W; European Uremic Toxin Work Group (EUTox). Review on uremic toxins: classification, concentration, and interindividual variability. Kidney Int. 2003 May;63(5):1934-43. doi: 10.1046/j.1523-1755.2003.00924.x. PMID 12675874
- [Background] Cohen G. Immunoglobulin light chains in uremia. Kidney Int Suppl. 2003 May;(84):S15-8. doi: 10.1046/j.1523-1755.63.s84.8.x. PMID 12694299
- [Background] Desjardins L, Liabeuf S, Lenglet A, Lemke HD, Vanholder R, Choukroun G, Massy ZA; European Uremic Toxin (EUTox) Work Group. Association between free light chain levels, and disease progression and mortality in chronic kidney disease. Toxins (Basel). 2013 Nov 8;5(11):2058-73. doi: 10.3390/toxins5112058. PMID 24217396
- [Background] Haynes R, Hutchison CA, Emberson J, Dasgupta T, Wheeler DC, Townend JN, Landray MJ, Cockwell P. Serum free light chains and the risk of ESRD and death in CKD. Clin J Am Soc Nephrol. 2011 Dec;6(12):2829-37. doi: 10.2215/CJN.03350411. Epub 2011 Oct 27. PMID 22034503
- [Background] Aoike I. Clinical significance of protein adsorbable membranes--long-term clinical effects and analysis using a proteomic technique. Nephrol Dial Transplant. 2007 Jul;22 Suppl 5:v13-9. doi: 10.1093/ndt/gfm295. PMID 17586841
- [Background] Hutchison CA, Blade J, Cockwell P, Cook M, Drayson M, Fermand JP, Kastritis E, Kyle R, Leung N, Pasquali S, Winearls C; International Kidney and Monoclonal Gammopathy Research Group. Novel approaches for reducing free light chains in patients with myeloma kidney. Nat Rev Nephrol. 2012 Feb 21;8(4):234-43. doi: 10.1038/nrneph.2012.14. PMID 22349488
- [Background] Testa A, Dejoie T, Lecarrer D, Wratten M, Sereni L, Renaux JL. Reduction of free immunoglobulin light chains using adsorption properties of hemodiafiltration with endogenous reinfusion. Blood Purif. 2010;30(1):34-6. doi: 10.1159/000316684. Epub 2010 Jun 24. PMID 20588010
- [Background] Borrelli S, Minutolo R, De Nicola L, De Simone E, De Simone W, Zito B, Guastaferro P, Nigro F, Iulianiello G, Credendino O, Bassi A, Leone L, Capuano M, Auricchio MR, Conte G. Effect of hemodiafiltration with endogenous reinfusion on overt idiopathic chronic inflammation in maintenance hemodialysis patients: a multicenter longitudinal study. Hemodial Int. 2014 Oct;18(4):758-66. doi: 10.1111/hdi.12178. Epub 2014 May 28. PMID 24865622
- [Background] Bourguignon C, Chenine L, Bargnoux AS, Leray-Moragues H, Canaud B, Cristol JP, Morena M. Hemodiafiltration improves free light chain removal and normalizes kappa/lambda ratio in hemodialysis patients. J Nephrol. 2016 Apr;29(2):251-257. doi: 10.1007/s40620-015-0207-z. Epub 2015 May 29. PMID 26022721
- [Background] Donati G, La Manna G, Cianciolo G, Grandinetti V, Carretta E, Cappuccilli M, Panicali L, Iorio M, Piscaglia F, Bolondi L, Coli L, Stefoni S. Extracorporeal detoxification for hepatic failure using molecular adsorbent recirculating system: depurative efficiency and clinical results in a long-term follow-up. Artif Organs. 2014 Feb;38(2):125-34. doi: 10.1111/aor.12106. Epub 2013 Jul 3. PMID 23834711
- [Background] Bergstrom J, Wehle B. No change in corrected beta 2-microglobulin concentration after cuprophane haemodialysis. Lancet. 1987 Mar 14;1(8533):628-9. doi: 10.1016/s0140-6736(87)90266-2. No abstract available. PMID 2881162
- [Background] Harding S, Provot F, Beuscart JB, Cook M, Bradwell AR, Stringer S, White D, Cockwell P, Hutchison CA. Aggregated serum free light chains may prevent adequate removal by high cut-off haemodialysis. Nephrol Dial Transplant. 2011 Apr;26(4):1438. doi: 10.1093/ndt/gfr019. Epub 2011 Mar 15. PMID 21406545
- [Background] Cohen G, Rudnicki M, Schmaldienst S, Horl WH. Effect of dialysis on serum/plasma levels of free immunoglobulin light chains in end-stage renal disease patients. Nephrol Dial Transplant. 2002 May;17(5):879-83. doi: 10.1093/ndt/17.5.879. PMID 11981077
- [Background] Fabbrini P, Sirtori S, Casiraghi E, Pieruzzi F, Genovesi S, Corti D, Brivio R, Gregorini G, Como G, Carati ML, Vigano MR, Stella A. Polymethylmethacrylate membrane and serum free light chain removal: enhancing adsorption properties. Blood Purif. 2013;35 Suppl 2:52-8. doi: 10.1159/000350849. Epub 2013 May 3. PMID 23676837
- [Background] Birk HW, Kistner A, Wizemann V, Schutterle G. Protein adsorption by artificial membrane materials under filtration conditions. Artif Organs. 1995 May;19(5):411-5. doi: 10.1111/j.1525-1594.1995.tb02351.x. PMID 7625919
- [Background] Lamy T, Henri P, Lobbedez T, Comby E, Ryckelynck JP, Ficheux M. Comparison between on-line high-efficiency hemodiafiltration and conventional high-flux hemodialysis for polyclonal free light chain removal. Blood Purif. 2014;37(2):93-8. doi: 10.1159/000357968. Epub 2014 Mar 1. PMID 24603634
- [Background] Stefoni S, Coli L, Cianciolo G, Donati G, Ruggeri G, Ramazzotti E, Pohlmeier R, Lang D. Inflammatory response of a new synthetic dialyzer membrane. A randomised cross-over comparison between polysulfone and helixone. Int J Artif Organs. 2003 Jan;26(1):26-32. doi: 10.1177/039139880302600105. PMID 12602466
- [Background] Rousseau-Gagnon M, Agharazii M, De Serres SA, Desmeules S. Effectiveness of Haemodiafiltration with Heat Sterilized High-Flux Polyphenylene HF Dialyzer in Reducing Free Light Chains in Patients with Myeloma Cast Nephropathy. PLoS One. 2015 Oct 14;10(10):e0140463. doi: 10.1371/journal.pone.0140463. eCollection 2015. PMID 26466100
- [Background] Cianciolo G, Coli L, La Manna G, Donati G, D'Addio F, Comai G, Ricci D, Dormi A, Wratten M, Feliciangeli G, Stefoni S. Is beta2-microglobulin-related amyloidosis of hemodialysis patients a multifactorial disease? A new pathogenetic approach. Int J Artif Organs. 2007 Oct;30(10):864-78. doi: 10.1177/039139880703001003. PMID 17992647
- [Background] Santoro A, Grazia M, Mancini E. The double polymethylmethacrylate filter (DELETE system) in the removal of light chains in chronic dialysis patients with multiple myeloma. Blood Purif. 2013;35 Suppl 2:5-13. doi: 10.1159/000350837. Epub 2013 May 3. PMID 23676829
- [Background] Pasquali S, Iannuzzella F, Corradini M, Mattei S, Bovino A, Stefani A, Palladino G, Caiazzo M. A novel option for reducing free light chains in myeloma kidney: supra-hemodiafiltration with endogenous reinfusion (HFR). J Nephrol. 2015 Apr;28(2):251-4. doi: 10.1007/s40620-014-0130-8. Epub 2014 Aug 23. PMID 25149172
- [Background] Machiguchi T, Tamura T, Yoshida H. Efficacy of haemodiafiltration treatment with PEPA dialysis membranes in plasma free light chain removal in a patient with primary amyloidosis. Nephrol Dial Transplant. 2002 Sep;17(9):1689-91. doi: 10.1093/ndt/17.9.1689. No abstract available. PMID 12198225
- [Derived] Donati G, Moretti MI, Baraldi O, Spazzoli A, Capelli I, Comai G, Marchetti A, Sarma M, Mancini R, La Manna G. Removal of free light chains in hemodialysis patients without multiple myeloma: a crossover comparison of three different dialyzers. BMC Nephrol. 2016 Nov 25;17(1):193. doi: 10.1186/s12882-016-0405-5. PMID 27884120